CLINICAL TRIAL: NCT06707415
Title: A Clinical Study to Compare the Accuracy and Precision of the MindTension Blink Eye Reflex Measuring (Evoked Response)Device to DANTAC Keypoint EMG System
Brief Title: Compare the Accuracy of MindTension Blink Eye Reflex Measuring Device to DANTAC Keypoint Electromyography (EMG) System.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MindTension (Industry)
Collaborators: Carmel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MND-03
Record Dates: First submitted 2024-09-18; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-06

CONDITIONS: Electromyography; Auditory Event-related Potential (AERP)
Keywords: MT1; Electromyography; Auditory evoked potentials
MeSH Terms: interventions — Evoked Potentials, Auditory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EMG evaluated group (Experimental): Participants are evaluated in both the MT1 and the Natus Dantec Keypoint systems
  Interventions: Diagnostic Test: Auditory evoked potentials

INTERVENTIONS:
Diagnostic Test: Auditory evoked potentials — Auditory evoked potentials in parallel systems

SUMMARY:
A clinical study aimed to compare the accuracy and precision of the MindTension MT1 auditory evoked response parallel to an FDA cleared device (Natus DANTEC Keypoint).

DETAILED DESCRIPTION:
Mindtension device measures the orbicularis muscle response to auditory stimuli, the device is backed up by an algorithm that calculates several parameters of startle reflex and startle related indices. In the present study we aim to test the validity, accuracy and precision of MT1 system compared to an FDA cleared device, the Natus DANTEC Keypoint EMG system (K944547).

The aim of this clinical trial is to demonstrate the accuracy and precision of the MT1 device to the FDA cleared Natus DANTEC Keypoint EMG system that is used in the EMG unit.

Participants (n=38) will be evaluated for eligibility of inclusion. As this is paired-group design study, patients will be randomized in a 1:1 ratio to group 1 (Right facial side with MT1 device), or group 2 (Right facial side Natus keypoint device), each patient will be tested using both devices at the same time. The test is 6 minutes in duration. The results will be compared within and between subject analysis.

Safety will be assessed through collection and analysis of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subject's informed consent.
* Healthy subjects, with no known chronic disease.
* Both genders, age between 18-45.

Exclusion Criteria:

* Any current co-morbid Chronic illness.
* Hearing loss.
* Pregnancy.
* Substance abuse during the last 3 months.
* Lack of cooperation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Average maximal peak levels | Day 1
  The average peak levels (in millivolts) following auditory stimulus.
Average peak index | Day 1
  The average index (in milliseconds) following auditory stimulus.
Average eye blink width | Day 1
  Average eye blink width (in milliseconds) following auditory stimuli.
Average inhibition | Day 1
  Average inhibition (in percent) following paired auditory stimuli.

SECONDARY OUTCOMES:
Average eye blink sum | Day 1
  Average eye blink sum (in millivolts) following auditory stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Shatz Azoulay, PhD, Study Director — MindTension
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No